CLINICAL TRIAL: NCT00722852
Title: Multicentre, Randomized, Double-blind, Placebo-controlled Study of Safety and Efficacy of Epicutaneously Applied Diractin® (Ketoprofen in Transfersome® Gel) for the Treatment of Osteoarthritis of the Knee
Brief Title: Study of Safety and Efficacy of Diractin® for the Treatment of Osteoarthritis (OA) of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IDEA AG (Industry)
Responsible Party: Dr. med. Matthias Rother, IDEA AG
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CL-033-III-06
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Last update posted 2009-10-05 (Estimated); Status verified 2009-10

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Ketoprofen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: ketoprofen in Diractin®
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ketoprofen in Diractin® — 100 mg (b.i.d.)
  Arms: 1
Drug: Placebo — 100 mg (b.i.d.)
  Arms: 2

SUMMARY:
The purpose of this study is to provide replicated evidence of safety and efficacy of 100 mg ketoprofen in Diractin®.

DETAILED DESCRIPTION:
The study will investigate safety and efficacy of Diractin® at relieving signs and symptoms of knee OA, including the primary endpoint of patient assessment of pain.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed and dated
* Age > 45 years
* Class I-III OA of the knee and subject meets American College of Rheumatology (ACR) clinical classification criteria for osteoarthritis of the knee

Exclusion Criteria:

* Skin lesions or dermatological diseases in the treatment area
* Directly or indirectly involved in the conduct and administration of this study
* Received any investigational medicinal product within 30 days prior to Screening Visit or participation in any previous clinical study with Diractin®
* Pregnancy or lactation
* Residents of psychiatric wards, prisons or other state institutions
* Malignancy within the past 2 years
* Depressive disorders requiring treatment with tricyclics, treatment with other antidepressants must be stable for 3 months prior to screening and throughout the study
* Epilepsy
* Schizophrenia
* Neuropathic pain and any other pain condition requiring chronic use of pain medication
* Known hypersensitivity or allergy (including photoallergy) to NSAID´s including ketoprofen and to ingredients of the IMP
* Preexisting asthma or bronchospasm after taking aspirin or other NSAIDs
* Unable to discontinue analgesic therapy including opioids, NSAID´s, tramadol, muscle relaxants, gabapentin, pregabalin, duloxetine, venlafaxine, capsaicine or other drugs approved or used for the treatment of pain for the duration of the study

Min Age: 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 555 (Actual)
Dates: Start 2008-06; Primary Completion 2009-02 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
pain subscale of the WOMAC | week 12

SECONDARY OUTCOMES:
Patient global assessment of response to therapy | week 12
function subscale of the WOMAC | week 12

CONTACTS AND LOCATIONS:
Overall Officials: IDEA AG, Study Director — IDEA AG
Locations (37):
- United States (37):
  - Hope Research Institute, Phoenix, Arizona
  - Premiere Pharmaceutical Research, Tempe, Arizona
  - Genova Clinical Research, Tucson, Arizona
  - Family Practice Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Orange County Clinical Trails, Inc., Anaheim, California
  - Encompass Clinical Research, Spring Valley, California
  - Tampa Bay Medical Research Inc., Clearwater, Florida
  - University Clinical Research DeLand, LCC, DeLand, Florida
  - Eastern Research, Hialeah, Florida
  - DSI, Jupiter, Florida
  - FPA Clinical Research, Kissimmee, Florida
  - Suncoast Clinical Research Family Practice, New Port Richey, Florida
  - Renstar Medical Research, Ocala, Florida
  - University Clinical Research, Inc., Pembroke Pines, Florida
  - Miami Research Associates, South Miami, Florida
  - Drug Studies America, Marietta, Georgia
  - Non-Surgical Orthopaedic & Spine Center, P.C., Marietta, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Advance Clinical Research Insititute, Boise, Idaho
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Integrated Clinical Trail Services, Inc., West Des Moines, Iowa
  - Lousianna Research Associates Inc. (LRC, Inc), New Orleans, Louisiana
  - Future Care Studies, Springfield, Massachusetts
  - Westside Family Medical Center, P.C., Kalamazoo, Michigan
  - Omaha Research, P.C., Omaha, Nebraska
  - Rochester Clinical Research, Rochester, New York
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - The Center of Clinical Research LLC, Winston-Salem, North Carolina
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Pharcotherapy Research Associate, Inc., Zanesville, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Founders Research Group Research, Philadelphia, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Coastal Carolina Research Center, Goose Creek, South Carolina
  - Sarah Cannon Research Institute, Jackson, Tennessee
  - Quality Research Inc., San Antonio, Texas
  - Progressive Clinical Research, San Antonio, Texas

REFERENCES:
- [Derived] Rother M, Conaghan PG. A randomized, double-blind, phase III trial in moderate osteoarthritis knee pain comparing topical ketoprofen gel with ketoprofen-free gel. J Rheumatol. 2013 Oct;40(10):1742-8. doi: 10.3899/jrheum.130192. Epub 2013 Sep 1. PMID 23996292